CLINICAL TRIAL: NCT02435017
Title: Nutrition Risk Screening in Chronic Kidney Disease (CKD) From the National Health and Nutrition Examination Survey
Brief Title: Dietary Phosphate and Serum Phosphorus
Status: Completed | Type: Observational
Sponsor: Linda W. Moore (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Linda W. Moore, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00001798
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Phosphorus Metabolism Disorders
Keywords: kidney disease; recommended dietary allowances; nutrition assessment; food; dietary proteins; Vitamin D; dietary fats; ethnology; Continental Population Groups; Phosphorus, dietary; Phosphorus/analysis
MeSH Terms: conditions — Phosphorus Metabolism Disorders; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults 20-85 years: Data from adults 20-85 years old will be evaluated for serum phosphorus concentration.

SUMMARY:
Overall study design is to review National Health and Nutrition Examination Survey (NHANES) data 1999-2008 for nutrition risk according to kidney function. Substudies will be performed to review the association of nutrients and overall dietary intake compared to biomarkers available in NHANES during this period.

DETAILED DESCRIPTION:
Data from NHANES 2003-2006 were used to evaluate the relationship between estimated dietary phosphorus intake and the measured serum phosphorus. The following variables were used:

1. Demographics: Age, sex, race/ethnicity
2. Dietary variables: Foods, food groups (as reported by the United States Department of Agriculture (USDA) method, further standardized to the Academy of Nutrition and Dietetics method for portion size and then divided into groups having inorganic phosphate additives or no inorganic phosphate additives), food weight (g), phosphorus (mg), dietary supplements
3. Socioeconomic variables: education, family income
4. Laboratory variables: serum creatinine, phosphorus; urine albumin, creatinine
5. Clinical assessments: hypertension (proportion having blood pressure ≥140 millimeters of mercury (mmHg) diastolic or ≥90 mmHg systolic or taking antihypertensive medications); hyperglycemia (proportion having serum glucose >126 mg/dL or taking medications for diabetes); kidney function based on Chronic Kidney Disease Epidemiology Collaboration (2009) equation, evaluated in 15 milliliters/min/1.73m2 increments from <15 to >105; anthropometrics (BMI, kg/m2; obesity class I, II, III)

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine

Exclusion Criteria:

* Pregnancy
* No dietary intake interview
* Dietary intake interview not valid
* Answered the question "Have you had dialysis in the past year?" as "Yes"

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the continuous NHANES program from 2003-2006 who met the inclusion/exclusion criteria were included in the analysis. NHANES samples the general US population to determine prevalence of major diseases and health risks by combining physical examination with laboratory studies and questionnaires in a standardized environment using trained personnel. Participants are selected through a complex, multistage, probability sampling approach.
Sampling Method: Probability Sample
Enrollment: 7895 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus concentration | approximately 24 hours
  Serum phosphorus concentration on the day that 24-hour dietary recall was obtained (reflecting dietary intake the day prior to blood draw); measured in mg/dL

SECONDARY OUTCOMES:
Kidney function level | Baseline
  Kidney function estimated from Chronic Kidney Disease Epidemiology Collaboration (2009) equation, mL/min/1.73m2, and separated into 15mL/min increments

CONTACTS AND LOCATIONS:
Overall Officials: Linda W Moore, MS, Principal Investigator — Director, Clinical Trials; Dept of Surgery

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] Moore LW, Byham-Gray LD, Scott Parrott J, Rigassio-Radler D, Mandayam S, Jones SL, Mitch WE, Osama Gaber A. The mean dietary protein intake at different stages of chronic kidney disease is higher than current guidelines. Kidney Int. 2013 Apr;83(4):724-32. doi: 10.1038/ki.2012.420. Epub 2013 Jan 9. PMID 23302719
- [Derived] Moore LW, Nolte JV, Gaber AO, Suki WN. Association of dietary phosphate and serum phosphorus concentration by levels of kidney function. Am J Clin Nutr. 2015 Aug;102(2):444-53. doi: 10.3945/ajcn.114.102715. Epub 2015 Jun 3. PMID 26040641